CLINICAL TRIAL: NCT03893929
Title: The Investigation of New Biological Markers for Prostate Cancer Diagnosis and Management in Chinese Population
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, NG Chi Fai, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2015.444
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chinese patients with clinical suspicious of prostate cancer: To identify potential new blood and urine markers for the diagnosis, risk stratification and prognosis prediction for prostate cancer in Chinese population.
  Interventions: Diagnostic Test: New Biological markers for prostate cancer diagnosis and management

INTERVENTIONS:
Diagnostic Test: New Biological markers for prostate cancer diagnosis and management — To identify potential new blood and urine markers for the diagnosis, risk stratification and prognosis prediction for prostate cancer in Chinese population.

SUMMARY:
Prostate cancer (PC) is highly prevalent worldwide and is currently the 3rd most commonly diagnosed prostate cancer in Hong Kong male population with more than 1600 new cases diagnosed per year. However, the current use of serum PSA as a diagnostic marker is unsatisfactory. Many patients has elevated serum PSA is actually due to other causes and also the level of serum PSA do not correlate with the staging and grading of prostate cancer. Moreover, the current risk stratification system, based on PSA, clinical staging and Gleason score is of only limited value, as a significant proportion of patients with high-risk nonmetastatic PC have incurable disease due to locally advanced and/or occult metastasis,, whilst others with indolent disease may never suffer morbidity or mortality from PC.

Therefore, in order to improve patient management and outcome, there is a need to identify newer markers and also validate some potential markers in Chinese population.

DETAILED DESCRIPTION:
Prostate cancer (PC) is highly prevalent worldwide and is currently the 3rd most commonly diagnosed prostate cancer in Hong Kong male population with more than 1600 new cases diagnosed per year. Even with widely used serum Prostate Specific Antigen (PSA) diagnostic testing, more than 50% men with newly diagnosed PC are deemed to have highrisk disease. 1 However, the current use of serum PSA as a diagnostic marker is unsatisfactory. Many patients has elevated serum PSA is actually due to other causes and also the level of serum PSA do not correlate with the staging and grading of prostate cancer. 2 Moreover, the current risk stratification system, based on PSA, clinical staging and Gleason score is of only limited value, as a significant proportion of patients with high-risk nonmetastatic PC have incurable disease due to locally advanced and/or occult metastasis, whilst others with indolent disease may never suffer morbidity or mortality from PC. Furthermore, high-risk (non-metastatic) prostate cancer (thus defined) exhibits a high degree of heterogeneity of response to current treatment protocols. Lastly, the characteristics of prostate cancer in our Chinese population might not be the same as those in Caucasian. 3,4 Several single biomarkers have been introduced in an attempt to address the clinical need for better prognostic tests in prostate cancer. For example, increased pre-operative PSA velocity (≥2ng/ml/per year) has been associated with increased risk of recurrence after prostatectomy5 and mortality6, as have increased serum levels of Kallikrein-2 and [-2]-pro PSA.7-10 Pre-operative levels of prostate cancer gene 3 (PCA3) have been found to be elevated in tumours >0.5cc, 11 however these findings could not be confirmed in recent work.12 Therefore, in order to improve patient management and outcome, there is therefore an urgent need to improve our ability to identify newer markers and also validate some potential markers in our population.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Chinese male patients with age > 18 years old
2. Clinical suspected to have prostate cancer, based on abnormal digital rectal examination or elevated serum PSA level

Exclusion Criteria:

1. Patient refused or unable to provide consent for the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 5000 Chinese patients with clinical suspicious of prostate cancer and pending for transrectal ultrasound (TRUS) guided prostate biopsy for assessment will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-10-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify potential new blood markers for the diagnosis for prostate cancer in Chinese population. | Baseline (One-time point)
  The application of Kallikrein-2 and [-2]-pro PSA in the diagnosis of prostate cancer in Chinese population.
To identify potential new blood markers for prognosis prediction for prostate cancer in Chinese population. | Baseline (One-time point)
  The application of Kallikrein-2 and [-2]-pro PSA in the prognosis of prostate cancer in Chinese population.
To identify potential new urine markers for the diagnosis for prostate cancer in Chinese population. | Baseline (One-time point)
  The role of urine spermine in the diagnosis of prostate cancer
To identify potential new urine markers for prognosis prediction for prostate cancer in Chinese population. | Baseline (One-time point)
  The role of urine spermine in the prognosis of prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ng CF, Chiu PK, Lam NY, Lam HC, Lee KW, Hou SS. The Prostate Health Index in predicting initial prostate biopsy outcomes in Asian men with prostate-specific antigen levels of 4-10 ng/mL. Int Urol Nephrol. 2014 Apr;46(4):711-7. doi: 10.1007/s11255-013-0582-0. Epub 2013 Oct 18. PMID 24136184
- [Background] Gudmundsson J, Sulem P, Gudbjartsson DF, Masson G, Agnarsson BA, Benediktsdottir KR, Sigurdsson A, Magnusson OT, Gudjonsson SA, Magnusdottir DN, Johannsdottir H, Helgadottir HT, Stacey SN, Jonasdottir A, Olafsdottir SB, Thorleifsson G, Jonasson JG, Tryggvadottir L, Navarrete S, Fuertes F, Helfand BT, Hu Q, Csiki IE, Mates IN, Jinga V, Aben KK, van Oort IM, Vermeulen SH, Donovan JL, Hamdy FC, Ng CF, Chiu PK, Lau KM, Ng MC, Gulcher JR, Kong A, Catalona WJ, Mayordomo JI, Einarsson GV, Barkardottir RB, Jonsson E, Mates D, Neal DE, Kiemeney LA, Thorsteinsdottir U, Rafnar T, Stefansson K. A study based on whole-genome sequencing yields a rare variant at 8q24 associated with prostate cancer. Nat Genet. 2012 Dec;44(12):1326-9. doi: 10.1038/ng.2437. Epub 2012 Oct 28. PMID 23104005
- [Background] Ren S, Peng Z, Mao JH, Yu Y, Yin C, Gao X, Cui Z, Zhang J, Yi K, Xu W, Chen C, Wang F, Guo X, Lu J, Yang J, Wei M, Tian Z, Guan Y, Tang L, Xu C, Wang L, Gao X, Tian W, Wang J, Yang H, Wang J, Sun Y. RNA-seq analysis of prostate cancer in the Chinese population identifies recurrent gene fusions, cancer-associated long noncoding RNAs and aberrant alternative splicings. Cell Res. 2012 May;22(5):806-21. doi: 10.1038/cr.2012.30. Epub 2012 Feb 21. PMID 22349460
- [Background] Patel DA, Presti JC Jr, McNeal JE, Gill H, Brooks JD, King CR. Preoperative PSA velocity is an independent prognostic factor for relapse after radical prostatectomy. J Clin Oncol. 2005 Sep 1;23(25):6157-62. doi: 10.1200/JCO.2005.01.2336. PMID 16135482
- [Background] D'Amico AV, Chen MH, Roehl KA, Catalona WJ. Preoperative PSA velocity and the risk of death from prostate cancer after radical prostatectomy. N Engl J Med. 2004 Jul 8;351(2):125-35. doi: 10.1056/NEJMoa032975. PMID 15247353
- [Background] Steuber T, Vickers AJ, Haese A, Becker C, Pettersson K, Chun FK, Kattan MW, Eastham JA, Scardino PT, Huland H, Lilja H. Risk assessment for biochemical recurrence prior to radical prostatectomy: significant enhancement contributed by human glandular kallikrein 2 (hK2) and free prostate specific antigen (PSA) in men with moderate PSA-elevation in serum. Int J Cancer. 2006 Mar 1;118(5):1234-40. doi: 10.1002/ijc.21474. PMID 16152616
- [Background] Haese A, Graefen M, Steuber T, Becker C, Pettersson K, Piironen T, Noldus J, Huland H, Lilja H. Human glandular kallikrein 2 levels in serum for discrimination of pathologically organ-confined from locally-advanced prostate cancer in total PSA-levels below 10 ng/ml. Prostate. 2001 Oct 1;49(2):101-9. doi: 10.1002/pros.1123. PMID 11582588
- [Background] Catalona WJ, Bartsch G, Rittenhouse HG, Evans CL, Linton HJ, Horninger W, Klocker H, Mikolajczyk SD. Serum pro-prostate specific antigen preferentially detects aggressive prostate cancers in men with 2 to 4 ng/ml prostate specific antigen. J Urol. 2004 Jun;171(6 Pt 1):2239-44. doi: 10.1097/01.ju.0000127737.94221.3e. PMID 15126794
- [Background] Stephan C, Kahrs AM, Cammann H, Lein M, Schrader M, Deger S, Miller K, Jung K. A [-2]proPSA-based artificial neural network significantly improves differentiation between prostate cancer and benign prostatic diseases. Prostate. 2009 Feb 1;69(2):198-207. doi: 10.1002/pros.20872. PMID 18942119
- [Background] Nakanishi H, Groskopf J, Fritsche HA, Bhadkamkar V, Blase A, Kumar SV, Davis JW, Troncoso P, Rittenhouse H, Babaian RJ. PCA3 molecular urine assay correlates with prostate cancer tumor volume: implication in selecting candidates for active surveillance. J Urol. 2008 May;179(5):1804-9; discussion 1809-10. doi: 10.1016/j.juro.2008.01.013. Epub 2008 Mar 18. PMID 18353398
- [Background] Hessels D, van Gils MP, van Hooij O, Jannink SA, Witjes JA, Verhaegh GW, Schalken JA. Predictive value of PCA3 in urinary sediments in determining clinico-pathological characteristics of prostate cancer. Prostate. 2010 Jan 1;70(1):10-6. doi: 10.1002/pros.21032. PMID 19708043
- [Background] Schipper RG, Romijn JC, Cuijpers VM, Verhofstad AA. Polyamines and prostatic cancer. Biochem Soc Trans. 2003 Apr;31(2):375-80. doi: 10.1042/bst0310375. PMID 12653642
- [Background] van der Graaf M, Schipper RG, Oosterhof GO, Schalken JA, Verhofstad AA, Heerschap A. Proton MR spectroscopy of prostatic tissue focused on the detection of spermine, a possible biomarker of malignant behavior in prostate cancer. MAGMA. 2000 Jul;10(3):153-9. doi: 10.1007/BF02590640. PMID 10873205